CLINICAL TRIAL: NCT05860322
Title: The Effect of Inulin Supplementation on Colonic Healing and Surgical Outcomes Following Colorectal Surgery
Brief Title: The Effect of Inulin Supplementation on Colorectal Surgery Outcomes
Acronym: INULINE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023-11342
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Anastomotic Complication
Keywords: colorectal cancer; inuline; anastomotic leak; anastomotic healing
MeSH Terms: conditions — Colorectal Neoplasms; Anastomotic Leak | interventions — Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inulin group (Experimental): Patients randomized to the intervention group will receive inulin supplementation for 14 days, preceding the surgery. Inulin will be given at a dosage of 10g/day divided in two doses.
  Interventions: Dietary Supplement: Inulin
- Control group (Placebo Comparator): Patients randomized to the control group will receive a placebo for 14 days, two times a day.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Inulin — Inulin is a water soluble non-digestible carbohydrate, and it is available in more than 36,000 species of plants. It is often used as dietary fiber and has obtained the "Generally recognized as safe" status (GRAS) by the Food and Drug Administration (FDA).
  Arms: Inulin group
Other: Placebo — Placebo control
  Arms: Control group

SUMMARY:
Colorectal cancer (CRC) is the third most diagnosed cancer in Canada. The most common surgical procedure in patients with CRC is an intestinal resection followed by a reconnection to rejoin the ends of the remaining bowel. Among the postoperative complications, leaking of this intestinal connection is notably feared, affecting up to 20% of patients. These leaks are characterized by impaired intestinal healing and are associated with severe infections and even death.

Various studies have shown that gut microbiota, the bacteria that live in the digestive tract, plays an essential role in intestinal healing following surgery. These results support the possibility of enhancing intestinal healing through supplements that act as an energy source for gut bacteria. Indeed, animal studies have shown that inulin supplementation, a fiber commonly found in plants, improves intestinal healing following bowel surgery. However, no studies in humans have evaluated its effects on CRC surgery patients.

This study aims to determine feasibility of a randomized controlled trial that assesses the effects of inulin supplementation before elective colorectal surgery.

DETAILED DESCRIPTION:
Based on preliminary data, our working hypotheses are that the gut microbiome plays a fundamental role in postoperative healing and that manipulation of preoperative microbiota using inulin will improve postoperative healing and prevent potential development of anastomotic leaks.

The pilot study aims to evaluate the feasibility of a randomized controlled trial that assesses the effects of inulin supplementation before elective colorectal surgery. The project has two main components, a clinical study, and a translational research. A randomized, multi-center, triple-blind, placebo-controlled clinical trial will be conducted to evaluate the impact of inulin supplementation on the clinical and oncological outcomes of inulin supplementation before elective colorectal oncological surgery. Mucosal, blood and fecal samples of patients with inulin supplementation will be compared with samples of patients without inulin supplementation.

The study objectives are:

1. Determine the tolerance of colorectal cancer patients to inulin supplementation before surgery.
2. Assess the effect of inulin supplementation on colonic healing and the rate of AL.
3. Determine the impact of inulin supplementation on the gut microbiota, the inflammatory markers, and the gut barrier function.
4. Assess the effect of inulin supplementation on CRC local and distant recurrence after surgery.

Identification of study participants

Patients who are about to undergo an oncological colorectal surgery will be recruited in the CHUM. Informed consent will be obtained from the patient before enrollment in the study.

Patients will be randomized to the inulin group (intervention group) or to the placebo group (control group). A stratified randomization will be conducted according to the sex (1- Male, 2-Female), the cancer location (1- Right and transverse colon, 2-Left colon and sigmoid, 3-Rectum) and the cancer grade.

Patients randomized to the intervention group will receive inulin supplementation for two weeks, preceding the surgery. Inulin will be given at a dosage of 10g/day divided in two doses. To foster compliance, the inulin will be provided in a calendar pill organizer. Patients randomized to the control group will receive a placebo for two weeks, twice a day. Placebo pills will be identical in appearance to the inulin pills. A total of 40 patients, 20 in each group, will be included in the pilot study.

Adequate colonic preparation will also be given to all the patients, including oral mechanical bowel preparation, oral antibiotics the day before surgery and intravenous antibiotics before surgical incision.

Collection of stool samples

Feces will be collected according to International Human Microbiome Standards (IHMS) guidelines (SOP 03). Two pre-operative specimens will be collected for each enrolled patient: pre-inulin/placebo supplementation and post-inulin/placebo supplementation.

Blood samples

Standard blood tests will be conducted for the participating patients. Supplementary volume will be collected during the per-operative test, before the surgery and at post-op day 3. Blood will be collected in two tubes to assess complete blood counts and to obtained serum.

Intraoperative mucosal sample

A mucosal biopsy coming from colonic anastomosis consist of a fragment from the transection line at the anastomosis. The specimen will be collected in a sterile tube and snap frozen.

Statistical Design

R, Stata and Prism will be used to perform the statistical analysis. Decision to use non-parametric tests is based on data normality (Shapiro-Wilk test) and homoscedasticity (Bartlett's test) tests. Multiple comparisons will be evaluated statistically by 1-way analysis of variance (ANOVA) or by Kruskal-Wallis test. Statistically significant differences will then be evaluated by two-tailed Student's t or Wilcoxon test. Multiple testing is corrected via False Discovery Rate estimation. For pre-supplementation and post-supplementation samples, a paired Student's t-test or paired Wilcoxon test will be used. For comparison of 2 groups, an unpaired Student's t-test or unpaired Wilcoxon test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a colorectal cancer and who present for elective colorectal surgery

Exclusion Criteria:

* Emergency surgery for perforation/obstruction.
* Use of antibiotics within 4 weeks prior to surgery (other than usual antibiotic prophylaxis).
* Presence of preoperative ileostomy or colostomy.
* Intestinal surgery within 4 weeks prior to colonic surgery.
* Active asthma.
* Presence of familial adenomatous polyposis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Gastrointestinal Symptom Rating Scale (GSRS) before and after treatment. | The questionnaires will be completed before treatment and after treatment (within the first week after surgery)
  The GSRS is a seven-point Likert-type scale with response options ranging from 1 (no discomfort at all) to 7 (very severe discomfort). It includes 15 questions that assess various gastrointestinal symptoms.
Change in the Digestion-associated Quality of Life Questionnaire (DQLQ) before and after treatment. | The questionnaires will be completed before treatment and after treatment (within the first week after surgery)
  The DQLQ is a 9-item questionnaire that uses a seven-point Likert-type scale to assess the impact of gastrointestinal symptoms on quality of life. The response options range from 'never' to 'always'.

SECONDARY OUTCOMES:
Anastomotic leak rate | Anastomotic leaks will be assessed clinically and, if needed, radiologically evaluated. The incidence of anastomotic leak will include cases that experience this complication during the first 12 weeks after surgery.
  All patients presenting with suspicious clinical features, such as worrisome laboratory results, post-operative fever, or abnormal physical examination findings, will undergo radiological examinations to confirm an anastomotic leak.
White blood cell count on post-operative day 3 | Blood sample will be collected on post-operative day 3.
  The white blood cell count will be monitored on post-operative day 3 to check for signs of infection or inflammation.
C-reactive protein (CRP) on post-operative day 3 | Blood sample will be collected on post-operative day 3.
  The CRP will be monitored on post-operative day 3 to check for signs of infection or inflammation.
Change in fecal calprotectin levels before treatment and after treatment (on the day before surgery). | Stool samples will be collected before treatment and after treatment (on the day before surgery)
  Changes in fecal calprotectin levels will be monitored to assess colonic inflammation.
MUC2 levels in the mucosal sample | The mucosal sample will be collected during surgery.
  MUC2 levels will assess the amount of mucin present in the mucosa, which is important for colonic healing after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carole Richard, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No